CLINICAL TRIAL: NCT02451397
Title: The Associations Analysis Between Lifestyle and Osteoporosis Among Chinese Population
Brief Title: Associations Analysis Between Lifestyle and Osteoporosis
Status: Completed | Type: Observational
Sponsor: Shanghai Tongji Hospital, Tongji University School of Medicine (Other)
Collaborators: Huashan Hospital (Other)
Responsible Party: Principal Investigator, Zihui Tang, M.D and Ph.D, Huashan Hospital
Other Study IDs: OPLA_Dr.Tang
Record Dates: First submitted 2015-04-13; First posted 2015-05-22 (Estimated); Last update posted 2021-01-06 (Actual); Status verified 2021-01

CONDITIONS: Osteoporosis of Disuse With Current Pathological Fracture

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Dr.Tang's research group: Chinese lifestyle associated with osteoporosis

INTERVENTIONS:
Other:  — This is a cross-sectional study, and we do not assign specific interventions to the subjects of the study.

SUMMARY:
A large-scale, community-based, cross-sectional study was conducted to evaluate the extent to which lifestyle was associated with osteoporosis among the Chinese population by using self-reported questionnaire methods.

DETAILED DESCRIPTION:
A large-scale, community-based, cross-sectional study was conducted to evaluate the extent to which lifestyle was associated with osteoporosis among the Chinese population by using self-reported questionnaire methods. More than 3000 participants were recruited in communities in Shanghai. Data involved in demographic information, lifestyle, dietary habits, medical history and clinical biomarkers were collected. Every participants were measured bone mineral density (BMD g/cm2) at calcaneus by standardized quantitative ultrasound (QUS, Hologic Inc., Bedford, MA, USA) utilizing T-scores based on WHO criteria. A standard statistical analysis including univariate and multiple variables regression analysis to explore the risk or preventive factors involved in Chinese lifestyle associated with osteoporosis.

ELIGIBILITY:
Inclusion Criteria:

* Participants aged 30-90 years were recruited from rural and urban communities in Shanghai.

Exclusion Criteria:

* Some participants with chronic diseases and conditions that might potentially affect bone mass, structure, or metabolism were excluded. Briefly, the exclusion criteria were as follows: a history of

  1. serious residual effects of cerebral vascular disease;
  2. serious chronic renal disease (Glomerular filtration rate - GFR < 30 mL/min/1.73m2);
  3. serious chronic liver disease or alcoholism;
  4. significant chronic lung disease;
  5. corticosteroid therapy at pharmacologic levels;
  6. evidence of other metabolic or inherited bone disease, such as hyper- or hypoparathyroidism, Paget disease, osteomalacia, or osteogenesis imperfecta;
  7. recent (within the past year) major gastrointestinal disease, such as peptic ulcer, malabsorption, chronic ulcerative colitis, regional enteritis, or significant chronic diarrhea;
  8. Cushing syndrome;
  9. hyperthyroidism; and
  10. any neurologic or musculoskeletal condition that would be a non-genetic cause of low bone mass.

Ages: 30 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: We performed a risk-factor study for osteoporosis using a random sample of the Chinese population. Participants were recruited from rural and urban communities in Shanghai. Survey participants aged 30-90 years were included in this study.
Sampling Method: Probability Sample
Enrollment: 3100 (Actual)
Dates: Start 2012-01 (Actual); Primary Completion 2018-08 (Actual); Study Completion 2020-12 (Actual)

PRIMARY OUTCOMES:
osteoporosis accessed by Bone Mass Density (BMD) | participants will be measured for the duration of outpatient stay, an expected average of 2 weeks
  The bone mineral density (BMD g/cm2) was measured at calcaneus by standardized quantitative ultrasound (QUS, Hologic Inc., Bedford, MA, USA) utilizing T-scores based on WHO criteria, which were obtained from the automated equipment. T-score refers to the ratio between patient's BMD and that of young adult population of same sex and ethnicity. T-score of > -1 was taken as normal, between -1 and -2.5 osteopenic and < -2.5 as osteoporotic.

CONTACTS AND LOCATIONS:
Overall Officials: Zihui Tang, M.D and Ph.D, Principal Investigator — Huashan Hospital
Locations (2):
- China (2):
  - Huasha Hospital, Shanghai, Shanghai Municipality
  - Huashan Hospital, Shanghai, Shanghai Municipality

REFERENCES:
- [Background] Tang ZH, Zeng F, Li Z, Zhou L. Association and predictive value analysis for resting heart rate and diabetes mellitus on cardiovascular autonomic neuropathy in general population. J Diabetes Res. 2014;2014:215473. doi: 10.1155/2014/215473. Epub 2014 Mar 18. PMID 24772443
- [Background] Tang ZH, Xiao P, Lei SF, Deng FY, Zhao LJ, Deng HY, Tan LJ, Shen H, Xiong DH, Recker RR, Deng HW. A bivariate whole-genome linkage scan suggests several shared genomic regions for obesity and osteoporosis. J Clin Endocrinol Metab. 2007 Jul;92(7):2751-7. doi: 10.1210/jc.2006-2607. Epub 2007 May 1. PMID 17473065
- [Background] Tang ZH, Wang L, Zeng F, Li Z, Yu X, Zhang K, Zhou L. Bayesian estimation of cardiovascular autonomic neuropathy diagnostic test based on short-term heart rate variability without a gold standard. BMJ Open. 2014 Oct 6;4(9):e005096. doi: 10.1136/bmjopen-2014-005096. PMID 25287103
- [Derived] Li X, Lei T, Tang Z, Dong J. Analyzing the association between fish consumption and osteoporosis in a sample of Chinese men. J Health Popul Nutr. 2017 Apr 19;36(1):13. doi: 10.1186/s41043-017-0088-y. PMID 28424092
- [Derived] Yu Q, Liu ZH, Lei T, Tang Z. Subjective evaluation of the frequency of coffee intake and relationship to osteoporosis in Chinese men. J Health Popul Nutr. 2016 Aug 5;35(1):24. doi: 10.1186/s41043-016-0060-2. PMID 27495290
- [Derived] Liu N, Zeng F, Zhang K, Tang Z. A community-based cross-sectional study for relationship of frequency of vegetables intake and osteoporosis in a Chinese postmenopausal women sample. BMC Womens Health. 2016 Jun 3;16:28. doi: 10.1186/s12905-016-0307-5. PMID 27259804
- [Derived] Yu CX, Zhang XZ, Zhang K, Tang Z. A cross-sectional study for estimation of associations between education level and osteoporosis in a Chinese men sample. BMC Musculoskelet Disord. 2015 Dec 9;16:382. doi: 10.1186/s12891-015-0839-0. PMID 26646811
- [Derived] Liu N, Chen J, Zhang K, Tang Z. A community-based study of the relationship between coronary artery disease and osteoporosis in Chinese postmenopausal women. Coron Artery Dis. 2016 Jan;27(1):59-64. doi: 10.1097/MCA.0000000000000306. PMID 26398152